CLINICAL TRIAL: NCT06578546
Title: A Single-arm, Open Label, Multicenter Clinical Study to Evaluate the Safety and Efficacy of VAO Regimen in Patients With Newly Diagnosed Ph-positive Acute Lymphoblastic Leukemia
Brief Title: Chemotherapy-free Regimen of Venetoclax, Azacitidine Plus Orebatinib (VAO Regimen) for Newly Diagnosed ph+ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAO
Record Dates: First submitted 2024-04-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-04

CONDITIONS: Ph-Positive Acute Lymphoblastic Leukemia
Keywords: Ph-positive ALL; Venetoclax+Azacitidine+Orebatinib
MeSH Terms: interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax, Azacitidine, and Orebatinib Regimen (Experimental): See Detailed Description.
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: Orebatinib

INTERVENTIONS:
Drug: Venetoclax — 100mg d1, 200mg d2, 400mg d2-21, oral (Adjusted according to the plasma concentration of venetoclax on day 4)，every 28 days for a treatment cycle.
Drug: Azacitidine — 75mg/m2 qd, d1-d7, subcutaneous injection, every 28 days for a treatment cycle.
Drug: Orebatinib — 20mg qod, d4-d21, oral, every 28 days for a treatment cycle.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Venetoclax, Azacitidine Plus Orebatinib in newly diagnosed Philadelphia chromosome-positive Acute Lymphoblastic Leukemia.

DETAILED DESCRIPTION:
This is a phase Ⅱ, single-arm, open Label, multicenter clinical study in newly diagnosed Ph-positive acute lymphoblastic leukemia patients. The patients will receive venetoclax, azacitidine and orebatinib regimen in the induction treatment. The patients who respond to induction treatment will undergo consolidation treatment, and an optional allogeneic hematopoietic stem cell transplantation and post-transplantation maintenance treatment with induction therapy according to patient's wishes.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed Ph-positive ALL without the history of chemotherapy or target therapy.
2. Age ≥18.
3. Eastern Cooperative Oncology Group (ECOG) score: 0-3.
4. Total serum bilirubin ≤ 2 x upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 1.5 x ULN, aspartate aminotransferase (AST) ≤ 1.5 x ULN.
5. Creatinine clearance ≥ 30 mL/min.
6. Serum lipase ≤ 1.5 x ULN, amylase =< 1.5 x ULN.
7. Provide informed consent.

Exclusion Criteria:

1. Patients with another malignant disease.
2. Patients with uncontrolled active infection.
3. Patients with left ventricular ejection fraction < 0.5 by echocardiography or grade III/IV cardiovascular dysfunction according to the New York Heart Association Classification.
4. Patients with HIV infection, active tuberculosis infection, or active hepatitis B or hepatitis C infection.
5. Patients with uncontrolled active bleeding.
6. Patients who has participated or participating in other clinical trials related to this disease.
7. Patients with history of previous chemotherapy or target therapy (except for oral hydroxyurea and/or leukopheresis for lowering white blood cell counts).
8. Pregnant and lactating women; patients of childbearing potential should be willing to practice methods of contraception throughout the study period.
9. Patients with other commodities that the investigators considered not suitable for the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
complete molecular remission（CMR） | End of cycle 1 and 2 (each cycle is 28 days)
  Proportion of patients achieving CMR at the end of 1 or 2 cycles

SECONDARY OUTCOMES:
CR | End of cycle 1 and 2 (each cycle is 28 days)
  Complete remission (CR) was defined as < 5% bone marrow blasts in an aspirate with spicules and independent of transfusions.
CRi | End of cycle 1 and 2 (each cycle is 28 days)
  CR with incomplete hematologic recovery (CRi) was defined as <5% bone marrow blasts, either ANC<1×10^9/L or platelets < 100×10^9/L, transfusion independence but with persistence of cytopenia.
MRD-negative CR | End of cycle 1 and 2 (each cycle is 28 days)
  Minimal residual disease (MRD)-negative CR was defined as a leukemic cell count below the sensitivity threshold of 1×10-4 (0.01%) bone marrow mononuclear cells (MNCs) by multiparameter flow cytometry.
CCyR | End of cycle 1 and 2 (each cycle is 28 days)
  Complete cytogenetic response (CCyR) was defined as lack of Ph in ≥ 20 bone marrow metaphases.
MMR | End of cycle 1 and 2 (each cycle is 28 days)
  Major molecular response (MMR) was defined as a BCR-ABL/ABL transcript ratio of 0.1% (international scale).
Number of adverse events | End of cycle 1 and 2 (each cycle is 28 days)
  Adverse events are evaluated with CTCAE V5.0
RFS | 1 year
  Relapse-free survival (RFS) was the duration from the day of CR to leukemia relapse, death, or last follow-up
OS | 1 year
  Overall survival (OS) was the time from enrollment to death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No